CLINICAL TRIAL: NCT06561360
Title: A Randomized, Multi-Center, Phase II Study of Vemurafenib Plus Obinutuzumab vs. Cladribine Plus Rituximab in Patients With Previously Untreated Hairy Cell Leukemia (HCL)
Brief Title: A Study of Vemurafenib and Obinutuzumab Compared to Cladribine and Rituximab in People With Hairy Cell Leukemia (HCL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-160
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Hairy Cell Leukemia
Keywords: Vemurafenib; Obinutuzumab; Cladribine; Rituximab; 24-160
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Vemurafenib; obinutuzumab; Cladribine; Rituximab

STUDY DESIGN:
Intervention Model Description: A randomized phase II multi-center, open-label, study of vemurafenib plus obinutuzumab (experimental arm) vs. cladribine plus rituximab (standard of care arm) in patients with previously untreated HCL.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vemurafenib plus Obinutuzumab (Experimental): Patients assigned to the study arm will receive vemurafenib orally twice daily (b.i.d.) continuously in cycles of 4 weeks (28 days) for a total of 4 cycles. Obinutuzumab will be administered concomitantly with vemurafenib starting at cycle 2 of treatment in cycles of 4 weeks. Obinutuzumab infusions will be administered on days 1, 8 and 15 during the cycle 2 and every 4 weeks during the cycle 3 and 4 of treatment.
  Interventions: Drug: Vemurafenib; Drug: Obinutuzumab
- Standard treatment of Cladribine plus Rituximab (Active Comparator): Patients assigned to the SOC arm will receive cladribine IV on days 1-5 concurrently with rituximab IV per week for 8 times, i.e., weekly x8 from day 1.
  Interventions: Drug: Cladribine; Drug: Rituximab

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib orally twice daily (b.i.d.) continuously in cycles of 4 weeks (28 days) for a total of 4 cycles.
  Arms: Vemurafenib plus Obinutuzumab
Drug: Obinutuzumab — Obinutuzumab will be administered concomitantly with vemurafenib starting at cycle 2 of treatment in cycles of 4 weeks.
  Arms: Vemurafenib plus Obinutuzumab
Drug: Cladribine — Cladribine IV on days 1-5 concurrently with rituximab.
  Arms: Standard treatment of Cladribine plus Rituximab
Drug: Rituximab — Rituximab on days 1-5 concurrently with rituximab.
  Arms: Standard treatment of Cladribine plus Rituximab

SUMMARY:
The researchers are doing this study to compare the safety of vemurafenib in combination with obinutuzumab to the standard of approach of cladribine in combination with rituximab. The researchers will look at which treatment causes fewer or milder side effects. Researchers think vemurafenib and obinutuzumab (non-chemotherapy drugs) may cause fewer side effects compared with the usual approach of chemotherapy drugs. They will also compare the two approaches to see which approach is more effective at eliminating cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age
* Histologically confirmed classical HCL by the enrolling institution
* Presence of BRAF V600E mutation as confirmed by PCR, NGS or immunohistochemistry. If patient is known to have negative BRAF mutation, repeat testing is advisable as well as discussion with the main study principal investigator.
* Has not received any prior therapy for the disease
* Patients who meet the standard treatment initiation criteria, as defined by ANC ≤1.0, Hgb ≤ 10.0 or PLT ≤100K
* ECOG performance status of 0 - 2
* Acceptable pre-study organ function during screening as defined as:

  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN; and
  * Serum creatinine ≤ 1.5x ULN
* Electrocardiogram (ECG) without evidence of clinically significant ventricular arrhythmias or ischemia as determined by the investigator and a rate-corrected QT interval (QTc, Bazett's formula) of < 480 msec
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of vemurafenib and cladribine, and 18 months after discontinuation of rituximab and obinutuzumab
* For men with female partners of childbearing potential, agreement to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of vemurafenib
* Negative serum pregnancy test within 7 days of commencement of treatment in women of childbearing potential

Exclusion Criteria:

* Have had previous treatment for HCL, including purine analogs, vemurafenib, rituximab, obinutuzumab, and other investigational agents. Previous treatment with transfusions and other supportive care such as G-CSF and erythropoietin are allowed.
* Known hypersensitivity to any of the study drugs.
* Patients with known long QT syndrome or uncorrectable electrolyte abnormalities
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibody

  ° Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing and take HBV viral prophylaxis such as entecavir.
* Known infection with HIV or human T-cell leukemia virus 1 (HTLV-1)
* Active uncontrolled infection, e.g. persistent bacteremia, supplemental oxygen or pressor supports, etc.
* Live vaccination within 28 days of randomization
* Patients with concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of the skin, in situ cervical cancer, adequately treated stage I/II cancer from which the patient is current in complete remission, or any other cancer from which the patient has been disease free for five years
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Patients with HCL variant (as defined by absence of expression of CD25)
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-09-09 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
incidences of ≥ grade 3 treatment-related toxicities | within 6 months of treatment
  per CTCAE v5.0 within first 6 months from the start of the treatment to account delayed toxicities of the treatments

SECONDARY OUTCOMES:
complete remission | 2 years
  Response will be determined by the Consensus Resolution response criteria.
  Complete response (CR)
  * A morphological absence of hairy cells in the blood and bone marrow
  * A normalization of any organomegaly and cytopenias
partial response | 2 years
  Partial response (PR)
  °A normalization of cytopenias
  °≥50% reduction in organomegaly and bone marrow hairy cells.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm